CLINICAL TRIAL: NCT04424017
Title: Sero-prevalence of Coronavirus Disease 2019 (COVID-19) in Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Egyptian Center for Research and Regenerative Medicine (Other Government)
Collaborators: Cairo University (Other); National Research Centre, Egypt (Other); Academy of Scientific Research and Technology, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19\004
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: COVID; Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthcare workers (HCWs)
  Interventions: Biological: Specific anti-SARS-CoV-2 antibodies
- Healthy blood donors and healthy subjects in blood bank
  Interventions: Biological: Specific anti-SARS-CoV-2 antibodies
- Convalescents
  Interventions: Biological: Specific anti-SARS-CoV-2 antibodies

INTERVENTIONS:
Biological: Specific anti-SARS-CoV-2 antibodies — A serum sample needs to be collected from each participant upon recruitment into the investigation All samples will be tested by the rapid test (Artron, Artron Laboratories, Burnaby, Canada), IgM / IgG which is an antibody capture Immunochromatografac assay for simultaneous detection of IgM and IgG in serum or plasma for COVID -19 in samples.
  All samples will be tested for total Immunoglobulins and IgG in samples for COVID-19 virus by Ortho clinical diagnostics chemiluminescent technique (Ortho, Raritan, USA).

SUMMARY:
The medical and paramedical staff of the front-line services are potentially exposed to SARS-CoV-2. Therefore, despite the application of standard protective measures, it is possible that a certain number of these personnel have already contracted SARS-CoV-2, including in its asymptomatic form. Serological testing in this context would be useful for deploying immune healthcare workers as to limit the risk of viral infection and transmission. Therefore, it is of utmost importance to prove that the serological response entails the production of neutralizing antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Not previously diagnosed with COVID-19 except for convalescents
* Not currently symptomatic with fever or respiratory symptoms (cough, dyspnea)

Exclusion Criteria:

* Patients with fever or respiratory symptoms (cough, dyspnea)
* Refusal to give informed consent, or contraindication to venipuncture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Age-stratified sample from general population with 3 subgroups:
  1. Healthcare workers (HCWs), comprising frontline doctors, nurses, health attendants, and receptionists.
  2. Healthy blood donors and healthy subjects in blood bank or laboratory (routine examinations as pre-employment, likely to be representative of the general population
  3. Convalescents
Sampling Method: Probability Sample
Enrollment: 1546 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Describe the serological status of individuals in the study by presence of specific anti-SARS-CoV-2 antibodies | 3 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - ECRRM, Cairo
  - Faculty of Medicine, Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No